CLINICAL TRIAL: NCT04278690
Title: A Randomized, Controlled Study of a Health Literacy-informed Technology-based Approach to Support Safe Medication Use by Parents After Discharge of Infants From the Neonatal Intensive Care Unit.
Brief Title: Supporting Safe Use of Medications by Parents After Infant Discharge From the Neonatal Intensive Care Unit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-01294
Record Dates: First submitted 2020-01-09; First posted 2020-02-20 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Medication Administered in Error

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Current usual care includes standard discharge counseling by a nurse, with or without additional MD counseling.
- HELPix (Experimental): HELPix parents will receive usual care as above, after which trained staff will generate HELPix patient-/regimen-specific medication instruction sheets and review them with the parent.
  Interventions: Other: HELPix
- HELPix+Tech (Experimental): After parent receives usual care and HELPix (as above), trained staff will walk parent through the app on-boarding process to overcome initial barriers to use. Steps: 1) Parent texted link to personalized on-line instructions. 2) Parent clicks link to app
  Interventions: Other: HELPix+Tech

INTERVENTIONS:
Other: HELPix — HELPix parents will receive usual care as above, after which trained staff will generate HELPix patient-/regimen-specific medication instruction sheets and review them with the parent. Instruction sheets include optimized instructions (mL-only, doses appropriately rounded, visuals of recommended tool (e.g. 1-mL syringe best for doses of <1 mL), explicit frequency information (e.g. 'morning and night' instead of '2x/day') reinforced by pictograms (e.g. sun/moon icons)). For each medication, staff will: 1) review the dose (refer to the pictographic dose diagram, which illustrates optimal dosing tool filled to correct amount), 2) demonstrate the dose using optimal dosing tool, 3) ask parent to 'teachback'/'showback' dose (e.g. parent shows provider how much they would give by pulling back plunger on syringe to right level), 4) provide optimal dosing tool for the parent to take home. We anticipate this process will take ~5-10 minutes.
  Arms: HELPix
Other: HELPix+Tech — After parent receives usual care and HELPix , trained staff will walk parent through the app on-boarding process to overcome initial barriers to use. Steps: 1) Parent texted link to personalized on-line instructions. 2) Parent clicks link to app. For each medicine: A. Dosing module with optimized instructions (c/w HELPix); parent teachback/showback of dose B. Frequency module supports simplified, explicit intervals (e.g. 'morning and night'), parent chooses convenient times (text reminders sent based on preferences). Time for TECH depends on # medicines and parent baseline knowledge; structured protocol used to see # teachback rounds needed .
  Arms: HELPix+Tech

SUMMARY:
This is a randomized controlled study of parents of children to be discharged from the neonatal intensive care unit at Bellevue and Elmhurst hospitals. A total of 425 subjects will be recruited across two sites over preparatory phases and two primary study phases.

DETAILED DESCRIPTION:
Our overarching goal is to promote safe medication use/adherence for high-risk infants, by leveraging health literacy approaches and mobile technology to reinforce provider counseling and support parent medication management after discharge from the NICU. We will adapt/integrate evidence-based strategies studied in less complex populations, for this vulnerable group. The HELPix (Health Education and Literacy for Parents) pictogram-based intervention, developed by our team, incorporates these strategies, with sizeable improvements found in medication knowledge, dosing errors, and adherence in outpatient general pediatric settings, but to date, HELPix has not been studied in NICU settings

ELIGIBILITY:
Inclusion Criteria:

1. English or Spanish-speaking
2. 18 years of age and older
3. Child discharged home with a Rx for >1 daily liquid medication (other than multivitamin)
4. Primary person who will administers child's medications.
5. Willingness and ability to participate

Exclusion Criteria:

1. Does not have a working phone number
2. Does not have access to internet (via computer/smartphone)
3. Does not have a mobile phone that receives texts.
4. Not able to return to the hospital for their child's follow-up visit
5. Visual acuity worse than 20/50 according to the Rosenbaum Pocket Screener
6. Uncorrectable hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Improvement in Dosing with HELPix+TECH and HELPix in comparison to usual care. | Visit 3 (Day 30)
  HELPix (health literacy-informed written materials and verbal counseling in addition to usual care) and HELPix+TECH (a health literacy-informed web application in addition to HELPix and usual care) will result in improved dosing compared to usual care alone. This will be assessed by the percentage of observed dosing error (whether clinically meaningful errors of >20% deviation and/or large error of >40% deviation).
Improvement in medication adherence with HELPix+TECH and HELPix in comparison to usual care | Visit 3 (Day 30)
  HELPix (health literacy-informed written materials and verbal counseling in addition to usual care) and HELPix+TECH (a health literacy-informed web application in addition to HELPix and usual care) will result in improved medication adherence compared to usual care alone. This will be assessed by the percentage of poor medication adherence (>20% deviation from # prescribed doses).

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang Sharon Yin, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request